CLINICAL TRIAL: NCT01850264
Title: Quartet™ Bad Oeynhausen Trial
Acronym: QUOTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Principal Investigator, Klaus Juergen Gutleben, Senior cardiologist, Heart and Diabetes Center North-Rhine Westfalia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HDZNRW_KA_002_KJG
Record Dates: First submitted 2012-12-19; First posted 2013-05-09 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Congestive Heart Failure; Cardiac Resynchronization Therapy
Keywords: cardiac resynchronization therapy; heart failure, congestive
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quadripolar LV electrode (Active Comparator): Application of a quadripolar LV electrode
  Interventions: Device: Application of quadripolar / bipolar LV electrodes
- Bipolar LV electrode (Active Comparator): Application of a bipolar LV electrode
  Interventions: Device: Application of quadripolar / bipolar LV electrodes

INTERVENTIONS:
Device: Application of quadripolar / bipolar LV electrodes

SUMMARY:
Primary objective of this study is to evaluate whether the use of a quadripolar left ventricular (LV) electrode compared to a standard bipolar LV electrode leads to lower non-responder rates in patients undergoing cardiac resynchronization therapy (CRT)

ELIGIBILITY:
Inclusion Criteria:

* Indication for CRT-D implantation according to current guidelines
* Ischemic cardiomyopathy (ICM) or dilated cardiomyopathy (DCM)
* Sinus rhythm
* NYHA II-IV
* Age ≥ 18 years
* Written informed consent to participate in the study

Exclusion Criteria:

* Right bundle brunch block
* Valvular cardiomyopathy
* Patient receiving a non-transvenous LV electrode
* Known pregnancy
* Age < 18 years
* Life expectancy < 1 year
* Atrial fibrillation / atrial flutter at the time of enrolment
* Inability to provide informed consent
* Participation in another study with active therapeutic arm
* Regular follow-up in the study center within the first 6 months after implantation not guaranteed

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-03; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Increase in peak oxygen consumption | 6 months
Reduction of New York Heart Association (NYHA) functional class | 6 months
Survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Klaus-Juergen Gutleben, M.D., Principal Investigator — Heart and Diabetes Center North Rhine-Westphalia, Department of Cardiology
Locations (1):
- Department of Cardiology, Heart and Diabetes Center North Rhine-Westphalia, Ruhr University Bochum, Bad Oeynhausen, Germany